CLINICAL TRIAL: NCT05804032
Title: A Randomized Phase III Non-inferiority Trial Assessing Lenalidomide, Bortezomib and Dexamethasone Induction Therapy with Either Intravenous or Subcutaneous Isatuximab in Transplant-eligible Patients with Newly Diagnosed Multiple Myeloma.
Brief Title: Lenalidomide, Bortezomib and Dexamethasone Induction Therapy with Either Intravenous or Subcutaneous Isatuximab in Patients with Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: Deutsche Studiengruppe Multiples Myelom (DSMM) (Unknown); KKS Netzwerk (Network); Sanofi (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Goldschmidt, Principal Investigator, University of Heidelberg Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMMG-HD8/DSMM XIX
Record Dates: First submitted 2023-03-21; First posted 2023-04-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Neoplasms; Paraproteinemias; Lymphoproliferative Disorders; Immunoproliferative Disorders; Lenalidomide; Bortezomib; Dexamethasone; Isatuximab; Monoclonal antibodies
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Paraproteinemias; Lymphoproliferative Disorders; Immunoproliferative Disorders | interventions — isatuximab; Lenalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - Intravenous isatuximab (Active Comparator): Patients in arm A are treated with 3 cycles RVd + i.v. isatuximab, followed by a standard intensification and autologous stem cell transplantation.
  Interventions: Drug: Isatuximab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone
- Arm B - Subcutaneous isatuximab (Experimental): Patients in arm B are treated with 3 cycles RVd + s.c. isatuximab, followed by a standard intensification and autologous stem cell transplantation.
  Interventions: Drug: Isatuximab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — IV isatuximab will be administered weekly in the first cycle (Cycle 1) on days 1, 8, 15, 22, 29, and biweekly on the 2 subsequent cycles at days 1, 15 and 29, at the dose of 10 mg/kg.
  Other Names: Sarclisa
  Arms: Arm A - Intravenous isatuximab
Drug: Isatuximab — SC isatuximab will be administered on days 1, 8, 15, 22, 29 of cycle 1, and on days 1, 15 and 29 of cycles 2-3, at the dose of 1400 mg
  Other Names: Sarclisa
  Arms: Arm B - Subcutaneous isatuximab
Drug: Lenalidomide — Both arms: 25 mg per os on day 1-14 and d22-35 in induction cycle 1-3
Drug: Bortezomib — Both arms: 1.3 mg/m^2 subcutaneous on day 1, 4, 8, 11, 22, 25, 29 32 in 3 induction cycles
  Other Names: Velcade
Drug: Dexamethasone — 20 mg per os on day 1-2, 4-5, 8-9, 11-12, 15; and 22-23, 25-26, 29-30, 32-33 in induction cycles 1-3.

SUMMARY:
The trial aims to demonstrate the non-inferiority of subcutaneous to intravenous isatuximab administration in transplant-eligible patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
Prospective, multicentre, randomised, parallel group, open, phase III clinical trial, for patients with confirmed diagnosis of untreated multiple myeloma requiring systemic therapy.

Investigational Medicinal Product: Isatuximab, subcutaneous administration via a wearable injector system.

Randomization: Patients are randomized in one of 2 study arms (A or B) before induction therapy. Patients randomized in arm A will receive 3 cycles of the monoclonal antibody isatuximab intravenously, combined with RVd regimen (Lenalidomide, Bortezomib, Dexamethasone). Each cycle will last for 42 days. Patients in arm B will receive 3 cycles RVd plus isatuximab subcutaneously. After induction therapy, patients will receive standard intensification (usually cyclophosphamide-based mobilization therapy, stem cell collection and high-dose melphalan followed by autologous stem cell transplantation (HDM/ASCT)). End of study will be after the first HDM/ASCT.

There is one primary objective:

Demonstration of non-inferiority of subcutaneous (SC) isatuximab compared to intravenous (IV) isatuximab, both in combination with RVd, with respect to rates of VGPR or better after induction therapy (according to standard International Myeloma Working Group (IMWG) response criteria).

Key secondary objectives are:

1. Comparison of patient-reported outcomes (PRO) regarding route of administration of isatuximab (SC vs. IV) on induction therapy as assessed by modified CTSQ (modified 9-item questionnaire).
2. Non-inferiority of rates of MRD negativity (assessed by NGS from BMA; sensitivity 10^-5) independent of standard IMWG response after induction therapy.

The duration of the trial for each patients is expected to be approximately 10 months (induction and intensification treatment).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of untreated MM requiring systemic therapy (diagnostic criteria according to IMWG)
* Patient is eligible for high-dose melphalan (200 mg/m^2 melphalan) and autologous stem cell transplantation
* Measurable MM disease according to IMWG criteria, defined as any quantifiable monoclonal protein value, defined by at least one of the following three measurements: serum M-protein ≥ 10 g/L; urine light-chain (M-protein) of ≥ 200 mg/24 hours; involved FLC level ≥ 10 mg/dL provided sFLC ratio is abnormal
* Age 18-70 years at trial inclusion

Exclusion Criteria:

* Patient has known hypersensitivity (or contraindication) to any of the components of study therapy
* Systemic amyloid light-chain amyloidosis (except for localized AL amyloidosis limited to the skin or the bone marrow)
* Plasma cell leukemia
* Previous chemotherapy or radiotherapy during the past 5 years except local radiotherapy in case of local MM progression
* Severe cardiac dysfunction (NYHA classification III-IV)
* Patients with active or uncontrolled hepatitis B or C or detectable liver disease due to hepatitis B or C
* HIV positivity
* Patients with active, uncontrolled infections
* Patients with severe renal insufficiency or requiring hemodialysis
* Patients with peripheral neuropathy or neuropathic pain, grade 2 or higher (as defined by the NCI Common Terminology Criteria for Adverse Events)
* Patients with a history of any active malignancy during the past 5 years with the exception of following malignancies after curative therapy: basal cell carcinoma of the skin, squamous cell skin carcinoma, stage 0 cervical carcinoma or any in situ malignancy
* Platelet count < 75 x 10^9/L
* Haemoglobin ≤ 8.0 g/dL, unless related to MM
* Absolute neutrophil count (ANC) < 1.0 x 10^9/L (the use of colony stimulating factors within 14 days before the test is not allowed)
* Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L)
* Pregnancy and lactation

For further details on inclusion/exclusion criteria please refer to the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-07-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Demonstration of non-inferiority of subcutaneous (SC) isatuximab compared to intravenous (IV) isatuximab, both in combination with RVd. | 18 weeks after start of study treatment
  Rates of VGPR or better (according to standard IMWG response criteria), defined as proportion of patients with at least VGPR after induction therapy (according to standard International Myeloma Working Group (IMWG) response criteria).

SECONDARY OUTCOMES:
Quality of life compared between Arm A and B. | 18 weeks after start of study treatment
  Comparison of PRO (patient-reported outcome) regarding route of administration of isatuximab (SC vs. IV) on induction therapy as assessed by modified CTSQ (modified 9-item questionnaire)
Non-inferiority of rates of MRD negativity in Arm B compared to Arm A | 18 weeks after start of study treatment
  Rates of NGS-MRD negativity (sensitivity 10^-5, from bone marrow aspirate) after induction therapy
Rates of MRD negativity by NGS and NGF (sensitivity 10^-5, from BMA) independent of standard IMWG response after first HDM/ASCT | 18 weeks (timepoint "after induction") or 35 weeks (timepoint "after first HDM/ASCT") after start of study treatment
  defined as proportion of negative patients with the corresponding MRD method (NGS or NGF) at the defined timepoint (after induction therapy or first HDM/ASCT)
Rates of best overall response to treatment (BOR) | Depending on the timepoint of best response out of all response assessments, up to 10 months from randomization
  proportion of patients with BOR (at least PR or better) to treatment until end of study (based on timepoints post induction cycle 2 and 3, prior to HDM/ASCT and post first HDM/ASCT)
Progression-free survival (PFS) | Until EOS (28 months after start of study)
  Time from randomization (at study inclusion) to progression or death from any cause whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Goldschmidt, Prof., Principal Investigator — GMMG study group
Locations (91):
- Austria (8):
  - Universitätsklinikum Krems, Krems
  - Ordensklinikum Linz, Linz
  - Landeskrankenhaus Feldkirch-Rankweil, Rankweil
  - Universitätsklinikum der Paracelsus, 3. Med. Abteilung/Onkologie Ambulanz, Salzburg
  - Universitätsklinikum St. Pölten - Lilienfeld, Sankt Pölten
  - Phyrn-Eisenwurzen Klinikum Steyr, Steyr
  - Klinik Ottakring, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Germany (83):
  - Uniklinik RWTH Aachen, Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzelltransplantation, Aachen
  - Asklepios Kliniken Hamburg GmbH, Altona
  - Klinikum Augsburg, II. Medizinische Klinik Hämatologie/Onkologie, Augsburg
  - Helios Klinikum Bad Saarow, Klinik für Hämatologie, Onkologie und Palliativmedizin, Bad Saarow
  - MedZentrum Klinikum Bayreuth GmbH, Bayreuth
  - Charité, III. Medizinische Abteilung (Hämatologie/Onkologie), Berlin
  - Vivantes Klinikum Neukölln, Klinik für Hämatologie und Onkologie, Berlin
  - Klinik für Hämatologie und Stammzelltransplantation, Helios Klinikum Berlin-Buch, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Bielefeld Praxis, Studiengesellschaft Onkologie, Bielefeld
  - Evangelisches Klinikum Bethel, Bielefeld
  - Johanniter-Krankenhaus Bonn, Bonn
  - Universitätsklinikum Bonn, Medizinische Klinik III, Bonn
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Carl-Thiem-Klinikum Cottbus gGmbH, 2. Medizinische Klinik, Cottbus
  - Klinikum Darmstadt, Medizinische Klinik V Hämatologie/Onkologie, Darmstadt
  - Städtisches Klinikum Dessau, Dessau
  - St.-Johannes-Hospital, Dortmund
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Medizinische Klinik und Poliklinik I, Dresden
  - Helios St. Johannes Klinik Duisburg, Medizinische Klinik 2, Duisburg
  - Universitätsklinikum Düsseldorf, Klinik für Hämatologie, Onkologie und Klinische Immunologie, Düsseldorf
  - Marien Hospital Düsseldorf GmbH, Klinik für Onkologie, Hämatalogie und Palliativmedizin, Düsseldorf
  - St. Antonius-Hospital Eschweiler, Klinik für Hämatologie / Onkologie, Eschweiler
  - Universitätsklinikum Essen, Essen
  - KEM I Evang. Kliniken Essen-Mitte gGmbH, Evangelisches Krankenhaus Essen-Werden gGmbH, Klinik für Hämatologie, Onkologie und Stammzelltransplantation, Essen
  - Malteser Krankenhaus, St. Franziskus Hospital, Hämatologie/Onkologie, Flensburg
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main
  - Universitätsklinikum Frankfurt, Medizinische Klinik 2, Hämatologie/Onkologie, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Gießen UK, Giessen
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Innere Medizin C, Greifswald
  - Katholisches Krankenhaus Hagen gGmbH, Klinik für Hämatologie und Onkologie, Hagen
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Zentrum für Onkologie, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Onkologische Schwerpunktpraxis Heidelberg, Heidelberg
  - Universitätsklinikum Heidelberg, Medizinische Klinik V, Heidelberg
  - SLK Kliniken Heilbronn, Medizinische Klinik III, Heilbronn
  - Universitätsklinikum des Saarlandes, Klinik für Innere Medizin 1, Homburg
  - Klinikum der Friedrich-Schiller-Universität Jena, Klinik für Innere Medizin II, Abteilung Hämatologie und internistische Onkologie, Jena
  - Westpfalz-Klinikum, Kaiserslautern
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikverbund Allgäu, Klinikum Kempten, Hämatologie / Onkologie, Kempten
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Gemeinschaftsklinikum Mittelrhein, Koblenz
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Lebach
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, III. Medizinische Klinik und Poliklinik, Mainz
  - Mannheimer Onkologie Praxis, Mannheim
  - Universitätsklinikum Mannheim, III. Medizinische Klinik, Mannheim
  - Philipps-Universität Marburg, Abteilung Hämatologie, Onkologie und Immunologie am Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Klinikum Hochsauerland, Meschede
  - Kliniken Maria Hilf GmbH, Medizinische Klinik I, Mönchengladbach
  - Kliniken Ostalb - Standort Stauferklinikum, Hämatologie und Onkologie, Mutlangen
  - Rotkreuzklinikum, München
  - Klinikum rechts der Isar der Technischen Universität München, Klinik und Poliklinik für Innere Medizin III, Hämatologie und Onkologie, München
  - Universitätsklinikum Münster, 1. Medizinische Klinik A, Münster
  - Klinikum Nürnberg, Nuremberg
  - Klinik Oldenburg, Oldenburg
  - Klinikum Osnabrück, Osnabrück
  - Brüderkrankenhaus St. Josef, Paderborn
  - Krankenhaus Barmherzige Brüder Regensburg, Klinik für Onkologie und Hämatologie, Regensburg
  - Universitätsklinikum Regensburg, Regensburg
  - CaritasKlinikum Saarbrücken St. Theresia, Saarbrücken
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Innere Medizin III (Tumorerkrankungen, Palliativmedizin), Schwäbisch Hall
  - Zentrum für ambulante Hämatologie und Onkologie (ZAHO), Siegburg
  - Onkologische Schwerpunktpraxis Speyer, Speyer
  - Klinikum der Landeshauptstadt Stuttgart - Katharinenhospital, Stuttgart
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universität Tübingen, Medizinische Universitätsklinik, Innere Medizin II: Onkologie, Hämatologie, Klinische Immunologie und Rheumatologie, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden GmbH, Wiesbaden
  - Helios Universitätsklinikum Wuppertal, Wuppertal
  - University of Würzburg, Med. Klinik und Poliklinik II, Würzburg

IPD SHARING:
Plan to Share IPD: No